CLINICAL TRIAL: NCT04848038
Title: Differential Effects of Exercise Modality on Cognition and Brain in Older Adults
Brief Title: Combined Exercise Trial
Acronym: COMET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 146904
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy Aging
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 1 of 4 study arms. Intervention arm include:
  1. core and fusion control condition;
  2. 150 minutes of endurance training (ET) only;
  3. 2 days a week of progressive weight training (WT) only;
  4. 150 minutes of ET and 2 days a week of WT.
  Participants exercise according to allocation for 1 year.
Who Masked: Outcomes Assessor
Masking Description: Raters (psychometrician, exercise physiologist) who perform outcome assessments will be blinded to the participant's intervention group. The study medical monitor and investigators will be unblinded to assist with safety assessments and address safety concerns or adverse events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Core and Fusion Training (Active Comparator): 150 minutes/week of Core and Fusion exercise, a mix of low impact toning, strengthening, flexibility and balance exercises.
  Interventions: Behavioral: Exercise
- Endurance Training (Active Comparator): Moderate-intensity endurance training such as brisk walking, 150 minutes/week over 3-5 days. Progression based on a set schedule. In addition 0-2 days of Core and Fusion control exercise will also be recommended.
  Interventions: Behavioral: Exercise
- Weight Training (Active Comparator): Progressive resistance training 2 days/week, non-consecutive, of 2 sets (10 - 15 repetitions) of 10 exercises (~75 minutes/week). Progression based on repetition completion and 1-repetition maximum. In addition 3 days of Core and Fusion control exercise will also be recommended.
  Interventions: Behavioral: Exercise
- Combined Endurance and Weight Training (Active Comparator): Moderate-intensity endurance training such as brisk walking, 150 minutes/week over 3-5 days. Progression based on a set schedule. Progressive resistance training 2 days/week, non-consecutive, of 2 sets (10 - 15 repetitions) of 10 exercises (~75 minutes/week). Progression based on repetition completion and 1-repetition maximum.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Standard public health exercise recommendations
  Other Names: Weight Training, Aerobic Exercise, Progressive Resistance Exercise, Cross Training

SUMMARY:
The number of older Americans will double in the next 4 decades to nearly 90 million, placing an unprecedented financial and resource burden on the health care system. Exercise has clear and demonstrable physical benefits, but a more precise understanding of how exercise supports cognitive function is essential. Demonstrating definitively that exercise as recommended by public health entities has benefits for cognition would have enormous public health implications, encourage the public to adapt more active lifestyles, and stimulate the development of effective exercise delivery programs.

DETAILED DESCRIPTION:
Older adults often experience physical decline that can be directly ameliorated by physical activity and exercise. Evidence is building that exercise prevents cognitive decline or delays the onset of debilitating dementia (e.g. Alzheimer's disease) yet, the optimal dose and combination of exercise modalities for promoting brain health, however, remains unknown and essentially untested.

The long-term research goal of this project is to develop and test strategies to support successful aging and prevent Alzheimer's disease. The study will enroll 280 individuals, age 65 to 80 years without cognitive impairment, into a 26-week exercise intervention to test the combined and independent effects of aerobic and resistance training on cognition, brain structure, and physical function. The project will also explore underlying biological mechanisms that may link exercise with brain health.

Participants will be randomized into 1 of 4 groups: flexibility, toning and balance (control), aerobic exercise training, progressive resistance training, or combined aerobic and resistance training. All intervention groups represent the most common modalities of exercise and directly reflect the public health recommendations for aerobic and resistance training. Exercise training will occur in a community setting through the network of Greater Kansas City Young Men's Christian Association. It is hypothesized that 26 weeks of exercise will improve 1) cognitive performance, 2) regional brain volume, 3) cardiorespiratory fitness and strength 4) biomarkers.

This will be the largest study to assess the combined and independent effects of the two most recommended forms of exercise. Demonstrating specific exercise effects on cognitive function and brain health in older adults would have enormous public health implications. The study's results will also impact public health policy and education by providing evidence towards the specific or synergistic effects of aerobic and resistance training on cognition and brain structure. Encouraging the public to adapt more active lifestyles and stimulate the development of effective exercise delivery programs to enhance initiation and maintenance of physical activity interventions is key to increasing the number of quality years of life for America's aging population.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-80 yrs (inclusive at time of consent).
* Conversant English speaking and reading ability.
* Medical clearance by a health care provider.
* Reliable means of transportation.
* Telephone Interview of Cognitive Status score > 25 and adjudication of normal cognition based on cognitive test data by a study medical monitor.

Exclusion Criteria:

* Intention to move out of the area or travel for more than 4 weeks in the next year.
* Use of an assistive device for ambulation.
* Joint pain severe enough to prevent taking walks in community, lifting objects over your head due to pain or restriction of movement, or that is worsened by increasing physical activity.
* Any MRI contraindications or refusal to attempt MRI.
* Treatment for alcohol or substance abuse in the last 2 years.
* Treatment for cancer (other than non-metastatic, localized cancer) in the last 2 years.
* Currently taking insulin.
* Diagnosis of heart disease, heart failure, heart attack, or heart surgery or chest pain with effort in the last 2 years.
* Untreated atrial fibrillation, valve replacements, angioplasty or stent placement in the last 2 years regardless of physician clearance.
* History of major psychiatric illness including schizophrenia (not including general anxiety disorder or depression), multiple sclerosis, Parkinson's, Dementia, mild cognitive impairment, brain injury (traumatic or clinically evident Stroke), or similar, likely to negatively impact cognitive testing.
* Head injury with loss of consciousness for more than a few minutes.
* Change in blood pressure medication in the last 2 months.
* Considered "Active" or engaging in a progressive resistance training 2 or more times a week.
* reported condition likely to compromise ability to safely perform exercise as determined by study medical monitor (e.g. chronic obstructive pulmonary disease, Lupus, end stage renal disease, etc.)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Global Cognition | Baseline, 6 months, 12 months
  Assessing change in cognitive function from baseline to 12 months. The 6 month measure is being used to assess the trajectory of the change. A comprehensive neuropsychological battery will be used that assesses a global cognition score derived from domains of cognition (e.g. Executive Function, Visuospatial Processing, Episodic Memory, Processing Speed). We will use a second order confirmatory factor analysis (CFA) to estimate the factor loadings between the observed indicators and the first order factors and between the first and second order factors. The CFA will use baseline data to avoid any potential intervention related biases. The primary outcome will be constructed by summing the weighted average (by the estimated first and second order loadings) of the standardized observed scores across the cognitive tests.

SECONDARY OUTCOMES:
Hippocampal volume | Baseline, 12 months
  Volume of bilateral hippocampus in milliliters
Peak oxygen consumption | Baseline, 12 months
  Peak volume of oxygen used in in milliliters per kilogram of body mass per minute during a graded maximal exercise test
1-Repetition Maximum | Baseline, 12 months
  The maximum amount of mass that can be lifted one time (summed leg press and chest press)

OTHER OUTCOMES:
Wechsler Test of Adult Reading | Baseline
  The Wechsler Test of Adult Reading is a reading recognition test that can be used to estimate intelligence quotient and memory scores
Hopkins Verbal Learning Test - Revised | Baseline, 6 months, 12 months
  The Hopkins Verbal Learning Test - Revised is an oral test that has been validated within brain-disordered populations (e.g., Alzheimer's disease, amnestic disorders) as a measure of verbal learning and memory.
NIH Toolbox Flanker Task | Baseline, 6 months, 12 months
  The NIH ToolboxFlanker Task is a computer based test to assess selective attention and inhibitory function.
NIH Toolbox Dimensional Change Card Sort | Baseline, 6 months, 12 months
  The NIH Toolbox Dimensional Change Card Sort is a computer based test to assess cognitive flexibility and attention.
NIH Toolbox Oral Symbol Digit Test | Baseline, 6 months, 12 months
  The NIH Toolbox Oral Symbol Digit Test is a computer based test to Measure of processing speed.
Virginia Cognitive Aging Project Logical Memory | Baseline, 6 months, 12 months
  The Virginia Cognitive Aging Project Logical Memory test measures episodic verbal memory.
Spatial Relations | Baseline, 26-weeks, 52-weeks
  In this computer task, participants are asked to determine which three-dimensional figure can be formed from a two-dimensional pattern presented. This task measures visual construction ability.
Letter Comparison | Baseline, 6 months, 12 months
  This paper-based task measures processing speed.
Matrix Reasoning | Baseline, 6 months, 12 months
  This computer-based task measures visuospatial ability.
Task Switching | Baseline, 6 months, 12 months
  This computer task asks participants to learn two different tasks. This task measures task switching.
Spatial Working Memory | Baseline, 6 months, 12 months
  This computer task measures spatial memory.
Stroop Task | Baseline, 6 months, 12 months
  This paper-based oral task measures executive control, specifically attention and inhibitory control.
Fat Mass | Baseline, 12 months
  Estimated total body, axial, appendicular and visceral fat mass from dual x-ray absorptiometry.
Lean Mass | Baseline, 12 months
  Estimated total body, axial, appendicular lean mass from dual x-ray absorptiometry.
Bone Mass | Baseline, 12 months
  Estimated total body, axial, appendicular bone mass and density from dual x-ray absorptiometry.
Cerebral brain blood flow | Baseline, 12 months
  Whole brain and regional cerebral blood flow estimated using arterial spin labeling, a technique of magnetic resonance imaging
Senior Fitness Test | Baseline, 12 months
  Composite and sub-test scores of 6 common physical activities. Scores can be normalized for age and sex
Waist to Hip Ratio | Baseline, 12 months
  The circumference of the waist and hip areas are measured via measuring tape.
Body Mass Index | Baseline, 12 months
  Height and body mass are measured and Body Mass Index is calculated based on a standard equation.
Blood lactate concentration | Baseline, 12 months
  Blood lactate concentration is measured before and after a bout of exercise.
MacArthur Scale of Subjective Social Status | Baseline, 6 months, 12 months
  The MacArthur Scale of Subjective Social Status (MacArthur Socio-Economic Status Scale) contains questions regarding finances, assets and other home socioeconomics.
Patient-Reported Outcomes Measurement Information System (PROMIS) Applied Cognitive Abilities v1.0 | Baseline, 6 months, 12 months
  Computer-based adaptive questionnaire of self-rated cognitive function.
Patient-Reported Outcomes Measurement Information System (PROMIS) Applied Cognitive General Concerns v1.0 | Baseline, 6 months, 12 months
  Computer-based adaptive questionnaire of self-rated cognitive concerns.
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety v1.0 | Baseline, 6 months, 12 months
  Computer-based adaptive questionnaire of self-rated anxiety.
Patient-Reported Outcomes Measurement Information System (PROMIS) Depression v1.0 | Baseline, 6 months, 12 months
  Computer-based adaptive questionnaire of self-rated depression.
Patient-Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities v1.0 | Baseline, 6 months, 12 months
  Computer-based adaptive questionnaire of self-rated social roles.
Patient-Reported Outcomes Measurement Information System (PROMIS) General Life Satisfaction v1.0 | Baseline, 6 months, 12 months
  Computer-based adaptive questionnaire of self-rated life satisfaction.
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function v1.0 | Baseline, 6 months, 12 months
  Computer-based adaptive questionnaire of self-rated life physical function.
Pittsburgh Sleep Quality Index | Baseline, 6 months, 12 months
  Paper-based questionnaire of self-rated sleep quality.
Perceived Stress Scale, 10-item | Baseline, 6 months, 12 months
  Paper-based questionnaire of self-rated appraisal of stress.
EuroQol Group Five Dimension Five Level (EQ-5D-5L) | Baseline, 6 months, 12 months
  A visual analog scale of quality of life
National Health and Nutrition Examination Survey Diet Survey Questionnaire | Baseline, 6 months, 12 months
  Self-rated computer based questionnaire of dietary intake.
Mediterranean Eating Pattern for Americans | Baseline, 6 months, 12 months
  Self-rated computer based questionnaire of mediterranean diet eating pattern.
Barriers Self-Efficacy Scale | Baseline, 3 months, 6 months, 12 months
  Self-rated computer based questionnaire of physical activity self-efficacy.
Exercise Self-Efficacy Scale | Baseline, 3 months, 6 months, 12 months
  Self-rated computer based questionnaire of exercise goal self-efficacy.
Leisure Self-Efficacy Scale | Baseline, 3 months, 6 months, 12 months
  Self-rated computer based questionnaire of leisure-time physical activity self-efficacy.
Physical Activity Self-Regulation Scale, 12-item | Baseline, 3 months, 6 months, 12 months
  Self-rated computer based measure of physical activity self-regulation for use with older adults.
Godin Leisure-Time Exercise Questionnaire | Baseline, 3 months, 6 months, 12 months
  Self-rated computer based measure of use of leisure-time for physical activity
Blood biomarkers | Baseline, 6 months, 12 months
  Brain Derived Neurotrophic factor , Insulin Growth Factor-1 (IGF-1), lactate, glucose and insulin levels, inflammatory cytokines, plasma phosphorylated tau (various form), plasma beta-amyloid (various forms), neurofilament light, glial fibrillary acidic protein and others as become available.

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Vidoni, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Alzheimer's Disease Center, Fairway, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
All data generated during the project will be entered into a secure database. This database will be housed on a secure network drive that is routinely backed-up to an offsite data storage location. Upon completion of the project, all data will be de-identified and available for other investigators at their request, in compliance with the NIH guidelines. It is not anticipated that unique resources will be developed and thus a plan for resource sharing is not provided.

REFERENCES:
- [Derived] Clutton J, Montgomery RN, Mudaranthakam DP, Blocker EM, Shaw AR, Szabo Reed AN, Vidoni ED. An open-source system for efficient clinical trial support: The COMET study experience. PLoS One. 2023 Nov 27;18(11):e0293874. doi: 10.1371/journal.pone.0293874. eCollection 2023. PMID 38011138